CLINICAL TRIAL: NCT04335578
Title: A Multicenter, Randomized, Placebo-Controlled Investigator-Blind, Participant-Blind Study to Evaluate Safety/Tolerability, Pharmacokinetics, and Pharmacodynamics of Zampilimab in Adult Kidney Transplant Recipients With Chronic Allograft Injury
Brief Title: A Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Zampilimab in Adult Kidney Transplant Recipients With Chronic Allograft Injury
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAI001; 2017-004807-31 (EudraCT Number)
Record Dates: First submitted 2020-04-03; First posted 2020-04-06 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Chronic Allograft Injury
Keywords: Chronic Allograft Injury; UCB7858; Kidney transplantation; CAI; zampilimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is an Investigator-blind and participant-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zampilimab Cohorts (Experimental): Participants will be randomized to receive zampilimab (UCB7858).
  Interventions: Drug: Zampilimab
- Placebo (Placebo Comparator): Participants randomized to this arm will receive matching Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zampilimab — Participants will receive zampilimab (UCB7858) at pre-specified time-points.
  Other Names: UCB7858
  Arms: Zampilimab Cohorts
Drug: Placebo — Participants will receive matching placebo (PBO) at pre-specified time-points.
  Other Names: PBO
  Arms: Placebo

SUMMARY:
The main purpose of the study is to investigate the safety and tolerability of repeat dosing with zampilimab in kidney transplant recipients with deteriorating kidney function associated with chronic allograft injury (CAI).

ELIGIBILITY:
Inclusion Criteria:

* Functioning living or deceased donor allograft >=1 year post-transplantation
* Baseline (screening) biopsy showing Grade II or III interstitial fibrosis/tubular atrophy (IF/TA) (>=25% IF/TA)
* Progressive loss in kidney function observed after the first year post-transplant, defined as an estimated glomerular filtration rate (eGFR) decline of ≥3 mL/min/year for at least 24 months prior to screening, with a minimum of 2 documented measurements per year (minimum of 4 documented measurements in the 24-month period, performed at least 1 month apart)
* An eGFR >=30 mL/min/1.73 m^2 for a period of 6 months up to screening
* Stable standard of care concomitant medication for 3 months prior to screening
* Participant is male or female, >=18 years of age

Exclusion Criteria:

* Recipient of multi-organ transplant (with the exception of repeated kidney transplant recipients, and/or corneal transplant recipients)
* Screening biopsy shows evidence of significant active antibody-mediated rejection that may affect the conduct of the study (eg, require change in treatment) according to the Principal Investigator (PI)
* Screening biopsy shows evidence of T cell-mediated rejection that may affect the conduct of the study (eg, require change in treatment) according to the PI
* Screening biopsy shows evidence of de novo or recurrent glomerular disease that may affect the conduct of the study (eg, require change in treatment) according to the PI
* Proteinuria ≥1500 mg/g at screening
* Participant who has a history of biopsy-proven acute rejection or treatment for suspected acute rejection within 3 months prior to screening
* Participant has had major surgery (including joint surgery) within 6 months prior to screening, or has planned surgery within 6 months after the last dose of investigational medicinal product (IMP)
* Participant has a current diagnosis of foot ulcer or diagnosis of chronic diabetic ulcer or history of delayed wound healing
* Participant has taken concomitant medication of sirolimus or everolimus within 3 months of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | From Day 1 (Baseline) to the end of Safety Follow-up Visit (up to Day 680)
  A treatment-emergent adverse event (TEAE) is defined as any event not present prior to the administration of investigational medicinal product (IMP) or any unresolved event already present before administration of IMP that worsens in intensity following exposure to the treatment.

SECONDARY OUTCOMES:
Serum concentration of zampilimab | From Day 1 (Baseline) to the end of Safety Follow-up Visit (up to Day 680)
  Serum concentration of the drug zampilimab from Baseline to the end of the last Safety Follow-up Visit
Urine concentration of zampilimab | From Day 1 (Baseline) to the end of Safety Follow-up Visit (up to Day 680)
  Urine concentration of the drug zampilimab from Baseline to the end of the last Safety Follow-up Visit

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Principal Investigator — 001 844 599 2273
Locations (5):
- Cai001 403, Nedlands, Australia
- Cai001 101, Leuven, Belgium
- Spain (2):
  - Cai001 301, Barcelona
  - Cai001 302, L'Hospitalet de Llobregat
- Cai001 501, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.

REFERENCES:
- [Derived] Zhou X, Trinh-Minh T, Matei AE, Gyorfi AH, Hong X, Bergmann C, Schett G, Atkinson J, Bowcutt R, Patel J, Johnson TS, Distler JHW. Amelioration of Fibrotic Remodeling of Human 3-Dimensional Full-Thickness Skin by Transglutamase 2 Inhibition. Arthritis Rheumatol. 2023 Sep;75(9):1619-1627. doi: 10.1002/art.42518. Epub 2023 Jul 5. PMID 37057394